CLINICAL TRIAL: NCT00002411
Title: A Randomized Study of the Long-Term Suppression of Plasma HIV RNA Levels by Triple Combination Regimens in Treatment Naive Subjects
Brief Title: A Comparison of Two Triple-Drug Combinations in Patients Who Have Never Been Treated With Anti-HIV Drugs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 039E; AI454-148
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2011-04-25 (Estimated); Status verified 2011-04

CONDITIONS: HIV Infections
Keywords: HIV-1; Didanosine; Drug Therapy, Combination; Zidovudine; Stavudine; Lamivudine; RNA, Viral; Nelfinavir; Anti-HIV Agents; Viral Load
MeSH Terms: conditions — HIV Infections | interventions — Nelfinavir; Lamivudine; Stavudine; Zidovudine; Didanosine

INTERVENTIONS:
Drug: Nelfinavir mesylate
Drug: Lamivudine
Drug: Stavudine
Drug: Zidovudine
Drug: Didanosine

SUMMARY:
The purpose of this study is to compare the safety of didanosine plus stavudine plus nelfinavir (NLF) with that of zidovudine plus lamivudine plus NLF. This study also examines how long these drug combinations are effective in lowering viral load (level of HIV in the blood).

ELIGIBILITY:
Inclusion Criteria

Patients must have:

Within 15 business days prior to randomization:

* CD4 cell count greater than or equal to 100 cells/mm3.
* HIV RNA greater than or equal to 2,000 copies/ml by Roche Amplicor Assay.

Exclusion Criteria

Co-existing Condition:

Patients with any of the following symptoms or conditions are excluded:

* Bilateral peripheral neuropathy.
* Intractable diarrhea.
* Proven or suspected acute hepatitis within 30 days prior to study entry.

Concurrent Medication:

Excluded:

- Therapy for any co-existing disease that may interfere with patient ability to participate in this study.

Concurrent Treatment:

Excluded:

Therapy for any co-existing disease that may interfere with patient ability to participate in this study.

Patients with the following prior conditions are excluded:

History of acute or chronic pancreatitis.

Prior Medication:

Excluded:

* Therapy for any previous disease that may interfere with patient ability to participate in this study.
* Excluded within 14 days prior to randomization:

Greater than 4 weeks of nucleoside therapy or greater than 1 week of protease inhibitor therapy.

* Excluded within 3 months of the start of this study or expected need at time of enrollment:
* Agents with significant systemic myelosuppressive, neurotoxic, pancreatoxic, hepatotoxic, or cytotoxic potential.
* Inability to tolerate oral medication.

Prior Treatment:

Excluded:

Therapy for any previous disease that may interfere with patient ability to participate in this study.

Risk Behavior:

Excluded:

Active alcohol or substance abuse that, in the opinion of the investigator, is sufficient to prevent adequate compliance with study therapy or to increase the risk of developing pancreatitis.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1998-03; Primary Completion 1999-09 (Actual); Study Completion 1999-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (32):
- United States (32):
  - Sorra Research Ctr / Med Forum, Birmingham, Alabama
  - Body Positive, Phoenix, Arizona
  - Hill Top Research Inc, Fresno, California
  - UCLA Med Ctr / CARE BH-412 CHS, Los Angeles, California
  - AIDS Healthcare Foundation, Los Angeles, California
  - West Los Angeles VAMC, Los Angeles, California
  - Sherman Oaks Hosp Research Institute, Sherman Oaks, California
  - Harbor UCLA Med Ctr / Research and Educational Institute, Torrance, California
  - Yale New Haven Hosp / Nathan Smith Clinic, New Haven, Connecticut
  - GW Med Ctr / Clinical Trials Unit, Washington D.C., District of Columbia
  - Med Alternatives, Fort Lauderdale, Florida
  - Urgent Care Ctr, Fort Lauderdale, Florida
  - Specialty Med Care Ctrs of South Florida Inc, Miami, Florida
  - Hillsborough County Health Dept, Tampa, Florida
  - Saint Josephs Hosp, Tampa, Florida
  - Northwestern Univ / Div of Infect Diseases, Chicago, Illinois
  - Rush Presbyterian / ST Lukes Med Ctr, Chicago, Illinois
  - Univ of Kansas School of Medicine / Office of Rsch, Wichita, Kansas
  - Ky Clinic Annex #4 / Room 205E / Speed Sort #0284, Lexington, Kentucky
  - Dartmouth-Hitchcock Med Ctr, Lebanon, New Hampshire
  - NJCRI, Newark, New Jersey
  - Infectious Disease Assoc of Central Jersey, Somerville, New Jersey
  - UCT International, Farmingdale, New York
  - St Luke Roosevelt Hosp, New York, New York
  - St Mary's Hosp (Univ of Rochester/Infectious Diseases), Rochester, New York
  - SUNY at Stony Brook / Div of Infectious Disease, Stony Brook, New York
  - Nalle Clinic / Clinical Research Dept, Charlotte, North Carolina
  - Associates in Med and Mental Health, Tulsa, Oklahoma
  - Stephen P Hauptman, Philadelphia, Pennsylvania
  - Med Univ of South Carolina / Div of Infect Disease, Charleston, South Carolina
  - Univ of Texas / Med Branch at Galveston, Galveston, Texas
  - Joseph C Gathe, Houston, Texas